CLINICAL TRIAL: NCT00939887
Title: A Phase 1, Healthy Volunteer Qualification Of Ligand [11C] PF-04767135 And Randomized Determination Of Kappa Opioid Receptor Occupancy Of PF-04455242, Using PET
Brief Title: A Study Of Kappa Opioid Receptor Occupancy Of PF-04455242, Using PET (Positron Emission Tomography)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: This study was terminated on January 6, 2010, due to toxicology findings in animals exposed to PF-04455242 for three months.
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Basic Science
Other Study IDs: B1071003
Record Dates: First submitted 2009-07-13; First posted 2009-07-15 (Estimated); Last update posted 2010-02-08 (Estimated); Status verified 2010-02

CONDITIONS: Bipolar Disorder; Depression
MeSH Terms: conditions — Bipolar Disorder; Depression | interventions — 2-methyl-N-((2'-(pyrrolidin-1-ylsulfonyl)biphenyl-4-yl)methyl)propan-1-amine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (Experimental)
  Interventions: Drug: PF-04455242

INTERVENTIONS:
Drug: PF-04455242 — Single dose of up to 30 mg PF-04455242, delivered in capsule.

SUMMARY:
This is a subject blind, investigator and sponsor open, randomized study consisting of 2 parts. Up to 15 healthy subjects will be included in the study. In the first part of the study the test retest reliability of the radiotracer [11C] PF 04767135 binding in man will be assessed. In the second part of this study, using [11C] PF 04767135, kappa opioid receptor occupancy (RO) will be assessed in up to three cohorts of subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female subjects of non-childbearing potential between the ages of 18 and 55 years, inclusive. (Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure and pulse rate measurement, 12 lead ECG and clinical laboratory tests.)

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing).
* Any condition possibly affecting drug absorption (eg, gastrectomy).
* A positive urine drug screen at Screening or Day 0.
* History of regular alcohol consumption exceeding 7 drinks/week for females or 14 drinks/week for men.
* Use of tobacco- or nicotine-containing products within 3 months of screening.
* Treatment with an investigational drug within 30 days or 5 half lives preceding the first dose of study medication (excluding [11C]PF 04767135).
* 12 lead ECG demonstrating QTc >450 msec at Screening.
* Pregnant or nursing females; females of childbearing potential.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2009-09; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Overall kappa opioid receptor occupancy of PF 04455242. | Study Day 1 and 2

SECONDARY OUTCOMES:
Binding potential (BP) of [11C] PF 04767135. | Study Day 1 and 2
Kappa opioid receptor occupancy of PF 04455242 at regions of interest in man. | Study Day 1 and 2
Relationship between plasma PF 04455242 concentration and kappa opioid receptor occupancy (IC50). | Study Day 1 and 2

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, New Haven, Connecticut, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1071003&StudyName=A%20Study%20Of%20Kappa%20Opioid%20Receptor%20Occupancy%20Of%20PF-04455242%2C%20Using%20PET%20%28Positron%20Emission%20Tomography%29